CLINICAL TRIAL: NCT06959771
Title: Base Editing Hematopoietic Stem Cell and BE T Cell Gene Therapy for CD40L-HyperIgM Syndrome-Single Patient Study
Brief Title: Base Editing Hematopoietic Stem Cell and T Cell Gene Therapy for CD40L-HyperIgM Syndrome: Single Patient Study
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10002385; 002385-I
Record Dates: First submitted 2025-05-06; First posted 2025-05-07 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12-29

CONDITIONS: CD40L-HyperIgM Syndrome
Keywords: base editing; Gene Editing
MeSH Terms: interventions — Alemtuzumab; Sirolimus; Fibroblast Growth Factor 7; Busulfan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm Study (Experimental): The study cell product is base edited autologous HSPCs which will be administered as a one-time infusion following conditioning using busulfan and alemtuzumab.
  Interventions: Biological: Base-edited hematopoietic stem and progenitor cells; Drug: Alemtuzumab; Drug: Sirolimus; Drug: Palifermin; Drug: Busulfan; Biological: Base-edited T lymphocyte cells

INTERVENTIONS:
Biological: Base-edited hematopoietic stem and progenitor cells — The study cell product is base edited autologous HSPCs which will be administered as a one-time infusion following myeloid conditioning.
Drug: Alemtuzumab — Serotherapy agent, 10 mg/m^2 on days -21, -20 and -19
Drug: Sirolimus — Immunophilin drug, will start on day -1, targeting a trough level between 4-12 ng/mL.
Drug: Palifermin — Mucositis prophylaxis agent, will be administered at 60 mcg/kg/day for 3 days before initiation of busulfan (days -6 to -4), as well as for the 3 days following study agent administration (days 1 to 3).
Drug: Busulfan — Myeloid conditioning agent, administered once daily (3 mg/kg) x 2 days, targeting a daily AUC of 4500 micromol*min/L or a cumulative AUC of 9000 micromol*min/L for the 2 days of therapy, if levels are available
Biological: Base-edited T lymphocyte cells — The secondary study cell product is base edited autologous which will be administered as a one-time infusion two weeks following the infusion of the base-edited autologous HSPCs.

SUMMARY:
Background:

X-linked hyper-IgM (HIGM) syndrome is caused by a mutation in the CD40 ligand (CD40L) gene. People with this disease have white blood cells that do not work properly. These people are at risk of severe infections and autoimmune diseases. Researchers want to know if these base-edited stem cells and T cells can help people with CD40L-HIGM syndrome.

Objective:

To test base-edited stem cells and base-edited T cells in 1 person with CD40L-HIGM syndrome.

Eligibility:

A single male with CD40L-HIGM syndrome.

Design:

A single participant is planned to receive a single dose of edited stem cells and supportive treatment with edited T cells. Participant stem and T cells will undergo base editing to repair the mutation.

In preparation for the gene therapy, the participant will receive busulfan chemotherapy and alemtuzumab. After treatment, the participant will have follow-up visits every few months in the first 2 years after treatment. Long-term visits will continue annually for 15 years.

DETAILED DESCRIPTION:
Study Description:

This is a single participant gene therapy study to provide a participant with CD40L c.658C>T; p.Q220X-Hyper IgM syndrome with autologous base-edited hematopoietic stem/progenitor cells (HSPC) and base-edited T cells (BE T). The study hypothesis is that base edited HSPCs will be repaired efficiently and safely to restore CD40L expression and improve immune function long term. BE T cells will provide functional T cells to support subject against immunodeficiency and lymphopenia.

The study cell product is base edited autologous HSPCs which will be administered as a one-time infusion following myeloid conditioning using busulfan administered once daily for 2 days with a daily target AUC of 4500 micromol*min/L or a cumulative AUC of 9000 micromol*min/L (approximately 6 mg/kg) and serotherapy (alemtuzumab (Campath)) 10 mg/m^2 total dose divided over 3 days by subcutaneous injection on days -21, -20, and -19. Following infusion, the participant will be evaluated at months 3, 6, 9, 12, 18, 24. Long-term annual follow up will be performed on a separate protocol.

Base edited autologous T cells will be administered at 2 weeks following BE HSPC infusion that function as 'donor lymphocyte infusions' to protect the patient from the diseaserelated T-cell immunodeficiency and alemtuzumab-related lymphopenia. Subsequent doses of BE T cells may be infused monthly as indicated to achieve T cell reconstitution for treatment of infections.

Objectives:

* Primary Objective: To determine the safety and efficacy of BE HSPC CD40L and BE T cells.
* Secondary Objectives: To determine restoration of CD40L expression and immune function
* Exploratory Objectives:

  * Assess for potential unintended edits
  * Kinetics of immune reconstitution

Endpoints:

* Primary Endpoint:

  * Efficacy determined by percentages of corrected alleles
  * Safety determined by toxicities related to infusion of Study Cell Product
* Secondary Endpoints:

  * Level of CD40L expression in peripheral blood T cells
  * IgG production
  * Response to immunization
* Exploratory Endpoints:

  * Repeat WES at 24 months after study cell product infusion
  * Evaluate for gene correction levels in peripheral blood CD34s and isolated immune cell lineages

ELIGIBILITY:
* INCLUSION CRITERIA:

This study is a single participant research study and to receive the study product, he needs to meet the following criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Has CD40L Q220X mutation
* Defective class switching
* Liver abnormalities (transaminases>UL)
* Portal hypertension
* Consensus from Hepatology Consult to receive myeloid conditioning
* Ability to take oral medication and be willing to adhere to the intervention regimen
* Use of condoms or other methods to ensure effective contraception with partner
* Ability of subject to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Known allergic reactions to components of the BE HSPC study product or BE T cell product
* Febrile illness within two weeks of hospital admission for treatment
* Unwilling to submit their information as part of the alemtuzumab (Campath(R)) Distribution Program application or the Distribution Program committee has determined the participant is not qualified to receive alemtuzumab.

NOTE: Alemtuzumab (campath) (IV formulation) is no longer distributed commercially. To receive product, the physician must contact the program for the participant. If the participant is not willing to consent to submit their info (demographics, contact information, and rationale for use) to the program such that we can obtain the drug, then we cannot proceed with conditioning; therefore no transplant will occur on this protocol. http://www.campath.com/

Co-enrollment guidelines: Co-enrollment in other trials is restricted, other than enrollment on observational studies and NIH protocols 94-I-0073 and 05-I-0213. Consideration for coenrollment in trials evaluating the use of a licensed medication will require the approval of the principal investigator in consultation with the medical monitor. Study staff should be notified of co-enrollment on any other protocol as it may require the approval of the principal investigator (in consultation with the medical monitor).

Ages: 37 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2027-10-28 (Estimated); Study Completion 2027-10-28 (Estimated)

PRIMARY OUTCOMES:
Safety determined by toxicities related to the infusion of the Study Cell Products | Through end of study
  To determine the safety and efficacy of BE HSPC CD40L and BE T Cells
Efficacy determined by percentages of corrected alleles | Through end of study
  To determine the safety and efficacy of BE HSPC CD40L and BE T Cells

SECONDARY OUTCOMES:
Level of CD40L expression in peripheral blood T cells | Through end of study
  To determine restoration of CD40L expression and immune function
IgG production | Through end of study
  To determine restoration of CD40L expression and immune function
Response to immunization | Through end of study
  To determine restoration of CD40L expression and immune function

CONTACTS AND LOCATIONS:
Overall Officials: Suk S De Ravin, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Winkelstein JA, Marino MC, Ochs H, Fuleihan R, Scholl PR, Geha R, Stiehm ER, Conley ME. The X-linked hyper-IgM syndrome: clinical and immunologic features of 79 patients. Medicine (Baltimore). 2003 Nov;82(6):373-84. doi: 10.1097/01.md.0000100046.06009.b0. PMID 14663287
- [Background] Kracker S, Gardes P, Durandy A. Inherited defects of immunoglobulin class switch recombination. Adv Exp Med Biol. 2010;685:166-74. doi: 10.1007/978-1-4419-6448-9_15. PMID 20687504
- [Background] Hubbard N, Hagin D, Sommer K, Song Y, Khan I, Clough C, Ochs HD, Rawlings DJ, Scharenberg AM, Torgerson TR. Targeted gene editing restores regulated CD40L function in X-linked hyper-IgM syndrome. Blood. 2016 May 26;127(21):2513-22. doi: 10.1182/blood-2015-11-683235. Epub 2016 Feb 22. PMID 26903548
- [Background] Ferrari S, Vavassori V, Canarutto D, Jacob A, Castiello MC, Javed AO, Genovese P. Gene Editing of Hematopoietic Stem Cells: Hopes and Hurdles Toward Clinical Translation. Front Genome Ed. 2021 Mar 31;3:618378. doi: 10.3389/fgeed.2021.618378. eCollection 2021. PMID 34713250
- [Background] Lazzarotto CR, Katta V, Li Y, Urbina E, Lee G, Tsai SQ. CHANGE-seq-BE enables simultaneously sensitive and unbiased in vitro profiling of base editor genome-wide activity. bioRxiv [Preprint]. 2024 Mar 30:2024.03.28.586621. doi: 10.1101/2024.03.28.586621. PMID 38585919
- [Background] de la Morena MT, Leonard D, Torgerson TR, Cabral-Marques O, Slatter M, Aghamohammadi A, Chandra S, Murguia-Favela L, Bonilla FA, Kanariou M, Damrongwatanasuk R, Kuo CY, Dvorak CC, Meyts I, Chen K, Kobrynski L, Kapoor N, Richter D, DiGiovanni D, Dhalla F, Farmaki E, Speckmann C, Espanol T, Shcherbina A, Hanson IC, Litzman J, Routes JM, Wong M, Fuleihan R, Seneviratne SL, Small TN, Janda A, Bezrodnik L, Seger R, Raccio AG, Edgar JD, Chou J, Abbott JK, van Montfrans J, Gonzalez-Granado LI, Bunin N, Kutukculer N, Gray P, Seminario G, Pasic S, Aquino V, Wysocki C, Abolhassani H, Dorsey M, Cunningham-Rundles C, Knutsen AP, Sleasman J, Costa Carvalho BT, Condino-Neto A, Grunebaum E, Chapel H, Ochs HD, Filipovich A, Cowan M, Gennery A, Cant A, Notarangelo LD, Roifman CM. Long-term outcomes of 176 patients with X-linked hyper-IgM syndrome treated with or without hematopoietic cell transplantation. J Allergy Clin Immunol. 2017 Apr;139(4):1282-1292. doi: 10.1016/j.jaci.2016.07.039. Epub 2016 Sep 30. PMID 27697500
- [Background] Gennery AR, Khawaja K, Veys P, Bredius RG, Notarangelo LD, Mazzolari E, Fischer A, Landais P, Cavazzana-Calvo M, Friedrich W, Fasth A, Wulffraat NM, Matthes-Martin S, Bensoussan D, Bordigoni P, Lange A, Pagliuca A, Andolina M, Cant AJ, Davies EG. Treatment of CD40 ligand deficiency by hematopoietic stem cell transplantation: a survey of the European experience, 1993-2002. Blood. 2004 Feb 1;103(3):1152-7. doi: 10.1182/blood-2003-06-2014. Epub 2003 Oct 2. PMID 14525761
- [Background] Vavassori V, Mercuri E, Marcovecchio GE, Castiello MC, Schiroli G, Albano L, Margulies C, Buquicchio F, Fontana E, Beretta S, Merelli I, Cappelleri A, Rancoita PM, Lougaris V, Plebani A, Kanariou M, Lankester A, Ferrua F, Scanziani E, Cotta-Ramusino C, Villa A, Naldini L, Genovese P. Modeling, optimization, and comparable efficacy of T cell and hematopoietic stem cell gene editing for treating hyper-IgM syndrome. EMBO Mol Med. 2021 Mar 5;13(3):e13545. doi: 10.15252/emmm.202013545. Epub 2021 Jan 21. PMID 33475257
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002385-I.html